CLINICAL TRIAL: NCT04352348
Title: Cohort of Patients Infected With SARS-CoV2 or Suspected of Being (COVID-19 in Ile-de-France)
Brief Title: Cohort of Patients Infected With SARS-CoV2 (COVID-19) or Suspected of Being
Acronym: COVIDeF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200382; 2020-A00754-35 (Other: ANSM)
Record Dates: First submitted 2020-03-31; First posted 2020-04-20 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: COVID-19; cohort; prognostic factors; severe forms
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COVID-19 negative (Other): Patients with exclusion diagnosis for COVID-19 infection
  Interventions: Other: blood samples; Other: feces samples (COVI-BIOME ancillary study); Other: sweat samples (COVIDOG ancillary study); Other: saliva samples; Other: Urine samples
- COVID-19 positive, not severe (Other): Patients with confirmed diagnosis of COVID-19 infection or suspected of being and not requiring hospitalization
  Interventions: Other: blood samples; Other: feces samples (COVI-BIOME ancillary study); Other: sweat samples (COVIDOG ancillary study); Other: saliva samples; Other: Phone call; Other: Urine samples
- COVID-19 positive, severe (Other): Patients with confirmed diagnosis of COVID-19 infection or suspected of being and requiring hospitalization
  Interventions: Other: blood samples; Other: feces samples (COVI-BIOME ancillary study); Other: sweat samples (COVIDOG ancillary study); Other: saliva samples; Other: 6 minutes walk test; Other: Phone call; Other: Urine samples
- Follow-up after COVID-19 hospitalization (Other): Patients previously hospitalized for COVID-19 infection but not recruited for the study can be recruited during a follow-up visit in hospital scheduled in standard care at 3 to 6 months after the hospitalization.
  For this arm, T0 = 3 to 6 months post-COVID-19 follow-up visit
  Interventions: Other: blood samples; Other: saliva samples; Other: 6 minutes walk test; Other: Phone call; Other: Urine samples

INTERVENTIONS:
Other: blood samples — All arms:
  1 blood sample at inclusion (T0)
  COVID-19 positive, severe only:
  1 blood sample at D3, at D7, in case of transfer to intensive care unit or in case of aggravation of symptoms, eventually, at discharge from hospital if the last blood sample was more than 3 days old, in case of post-COVID-19 follow-up visit scheduled in standard care at 3 to 6 months after hospitalization and in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization.
  Follow-up after COVID-19 hospitalization only:
  1 blood sample in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization
Other: feces samples (COVI-BIOME ancillary study) — All arms:
  1 feces sample at inclusion (T0)
  COVID-19 positive, severe only:
  1 feces sample at D3, at D7, in case of transfer to intensive care unit or in case of aggravation of symptoms and, eventually, at discharge from hospital
  Arms: COVID-19 negative; COVID-19 positive, not severe; COVID-19 positive, severe
Other: sweat samples (COVIDOG ancillary study) — All arms:
  2 sweat samples at inclusion (T0)
  Arms: COVID-19 negative; COVID-19 positive, not severe; COVID-19 positive, severe
Other: saliva samples — All arms:
  1 saliva sample at inclusion (T0)
  COVID-19 positive, severe only:
  1 saliva sample at D7, at discharge from hospital, in case of post-COVID-19 follow-up visit scheduled in standard care at 3 to 6 months after hospitalization and in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization.
  Follow-up after COVID-19 hospitalization only:
  1 blood sample in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization
Other: 6 minutes walk test — COVID-19 positive, severe only:
  6 minutes walk test in case of post-COVID-19 follow-up visit scheduled in standard care at 3 to 6 months after hospitalization and in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization.
  Follow-up after COVID-19 hospitalization only:
  6 minutes walk test at inclusion (T0) and in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization.
  Arms: COVID-19 positive, severe; Follow-up after COVID-19 hospitalization
Other: Phone call — All arms except COVID-19 negative:
  1 phone call 3 months after COVID-19 infection.
  All arms except COVID-19 negative:
  1 phone call 6 months after COVID-19 infection.
  All arms except COVID-19 negative:
  1 phone call 12 months after COVID-19 infection.
  Arms: COVID-19 positive, not severe; COVID-19 positive, severe; Follow-up after COVID-19 hospitalization
Other: Urine samples — All arms:
  1 urine sample at inclusion (T0)
  COVID-19 positive, severe only:
  1 urine sample at D3, at D7, at discharge from hospital, in case of post-COVID-19 follow-up visit scheduled in standard care at 3 to 6 months after hospitalization and in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization.
  Follow-up after COVID-19 hospitalization only:
  1 urine sample in case of post-COVID-19 follow-up visit scheduled in standard care at 11 to 13 months after hospitalization

SUMMARY:
On 17th March 2020, 198 193 confirmed cases (7 730 in France) of COVID-19 infections and 7 854 deaths (175 in France) have been reported from 8th December 2019 in 157 countries. The rapid increase in cases on french territory has led to the transition of France to level 3 of the epidemic on 14th March 2020.

The natural history of the disease is still poorly understood, especially prognostic factors, which are crucial for the best medical care of patients in times of epidemics, when hospital capacities are under pressure.

A better knowledge of natural history, of prognostic factors, the development and validation of new diagnostic tests, the evaluation of medical care, will lead to a better medical care of patients infected with COVID-19.

DETAILED DESCRIPTION:
The principal goal of the research is to assess the prognostic factors of the progression toward severe forms of the COVID-19 infection.

The secondary aims of the study are to contribute to answer some of the WHO research priority goals on COVID-19 infections:

* description of the natural history of the disease, its different forms, its clinical characterisation, its progression profile, the natural history of the disease linked to patient profiles
* evaluation and to comparison of different diagnostic methods, linked to the medical case
* description of the progression of the immune response during the infection and related to its outcome
* description of the replication and the excretion of the virus
* description of the progression of the biological markers during the infection and related to its outcome
* identification of the prognostic factors of the evolutive profile, especially if negative
* description of the patients care
* evaluation of the impact of the different therapeutic managements on the clinical outcome, the immune response, the viral load and the biomarkers.
* modeling of the epidemiologic impact
* identification of targets for treatment development
* analysis of cost data linked to the progression The population will include all patients infected with SARS-CoV2 ou suspected of being, who are taken care of at hospital.

The research is based on the collection of clinical and biological data from routine cares and on the biological analysis of blood samples.

The principal goal of the COVI-BIOME ancillary study is to identify gastrointestinal predictive factors for a severe form of the COVID-19 infection.

The principal goal of the COVIDOG ancillary study is to evaluate the sensibility and the specificity of canine olfactory detection for the volatile organic compounds of SARS-CoV2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patient admitted in an emergency unit or hospitalized, infected with SARS-CoV2 or suspected of being (the recruitment can occured during acute episode or during a follow-up visit)
* Written informed consent or emergency procedure
* Affiliated to health insurance system

Exclusion Criteria:

* Refusal of participation
* Patient under justice protection measure except guardianship and trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2003 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Identification of prognostic factors for progression to a severe form of COVID-19 infection | 12 months
  Research of prognostic factors which could be implicated in the progression to severe form of COVID-19 infection.

SECONDARY OUTCOMES:
Clinical aggravation of the infection | 12 months
Discharge of hospitalization | 12 months
Death | 12 months
Description of clinical manifestations | 12 months
Description of biological manifestations | 12 months
Description of radiological manifestations | 12 months
Description of physiological manifestations | 12 months
Patient-related prognostic factors | 12 months
Virus-related risk factors | 12 months
Comparison of the results of different diagnosis tests | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre HAUSFATER, MD, Principal Investigator — GH Pitié Salpêtrière - Charles Foix
Locations (1):
- GH Pitié-Salpêtrière / Service d'Accueil des Urgences, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cancella de Abreu M, Ropers J, Oueidat N, Pieroni L, Frere C, Fontenay M, Torelino K, Chauvin A, Hekimian G, Marcelin AG, Parfait B, Tubach F, Hausfater P; COVIDeF study group. Biomarkers of COVID-19 short-term worsening: a multiparameter analysis within the prospective multicenter COVIDeF cohort. Eur J Emerg Med. 2024 Dec 1;31(6):429-437. doi: 10.1097/MEJ.0000000000001175. Epub 2024 Sep 12. PMID 39480645
- [Derived] Matuozzo D, Talouarn E, Marchal A, Zhang P, Manry J, Seeleuthner Y, Zhang Y, Bolze A, Chaldebas M, Milisavljevic B, Gervais A, Bastard P, Asano T, Bizien L, Barzaghi F, Abolhassani H, Abou Tayoun A, Aiuti A, Alavi Darazam I, Allende LM, Alonso-Arias R, Arias AA, Aytekin G, Bergman P, Bondesan S, Bryceson YT, Bustos IG, Cabrera-Marante O, Carcel S, Carrera P, Casari G, Chaibi K, Colobran R, Condino-Neto A, Covill LE, Delmonte OM, El Zein L, Flores C, Gregersen PK, Gut M, Haerynck F, Halwani R, Hancerli S, Hammarstrom L, Hatipoglu N, Karbuz A, Keles S, Kyheng C, Leon-Lopez R, Franco JL, Mansouri D, Martinez-Picado J, Metin Akcan O, Migeotte I, Morange PE, Morelle G, Martin-Nalda A, Novelli G, Novelli A, Ozcelik T, Palabiyik F, Pan-Hammarstrom Q, de Diego RP, Planas-Serra L, Pleguezuelo DE, Prando C, Pujol A, Reyes LF, Riviere JG, Rodriguez-Gallego C, Rojas J, Rovere-Querini P, Schluter A, Shahrooei M, Sobh A, Soler-Palacin P, Tandjaoui-Lambiotte Y, Tipu I, Tresoldi C, Troya J, van de Beek D, Zatz M, Zawadzki P, Al-Muhsen SZ, Alosaimi MF, Alsohime FM, Baris-Feldman H, Butte MJ, Constantinescu SN, Cooper MA, Dalgard CL, Fellay J, Heath JR, Lau YL, Lifton RP, Maniatis T, Mogensen TH, von Bernuth H, Lermine A, Vidaud M, Boland A, Deleuze JF, Nussbaum R, Kahn-Kirby A, Mentre F, Tubiana S, Gorochov G, Tubach F, Hausfater P; COVID Human Genetic Effort; COVIDeF Study Group; French COVID Cohort Study Group; CoV-Contact Cohort; COVID-STORM Clinicians; COVID Clinicians; Orchestra Working Group; Amsterdam UMC Covid-19 Biobank; NIAID-USUHS COVID Study Group; Meyts I, Zhang SY, Puel A, Notarangelo LD, Boisson-Dupuis S, Su HC, Boisson B, Jouanguy E, Casanova JL, Zhang Q, Abel L, Cobat A. Rare predicted loss-of-function variants of type I IFN immunity genes are associated with life-threatening COVID-19. Genome Med. 2023 Apr 5;15(1):22. doi: 10.1186/s13073-023-01173-8. PMID 37020259